CLINICAL TRIAL: NCT04475237
Title: Virtual Anatomical Reconstruction of Mandibular Bone Defects Using a Statistical Shape Model
Status: Completed | Type: Observational
Sponsor: CADskills (Industry)
Responsible Party: Sponsor
Other Study IDs: SSM
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Mandibular Diseases; SSM
MeSH Terms: conditions — Mandibular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy mandibles: Belgian adults (between 20 and 60 years old), 50/50 male/female, with no major mandibular problems/deformities
  Interventions: Other: CT-scan evaluation and segmentation

INTERVENTIONS:
Other: CT-scan evaluation and segmentation — CT-scans will be evaluated (to see if they are included in the research group) and segmented if they are accepted.

SUMMARY:
Hundred already taken CT-scans (50 male and 50 female) will be anonymized. These scans will be segmented and implemented into a statistical shape model that will be used to predict missing hard tissue of a mandible based on the remaining bone.

DETAILED DESCRIPTION:
Together with the radiology and Craniomaxillofacial (CMF) department, 100 scans will be selected from the database (50 males and 50 females, between 20 and 60 years old). First, they will be anonymized (except the sex and age/date of birth). Afterwards, they will be segmented using Materialise Mimics software. The segmented mandibles will then be used to create a statistical shape model (SSM) using principal component analysis. This model will afterwards be used to predict the mandibular shapes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mandibles

Exclusion Criteria:

* Mandibles with major deformities
* Mandibles with obvious problems
* Mandibles that already underwent surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: European adults
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
A statistical shape model of a mandible | 2 months
  A statistical shape model of a mandible

CONTACTS AND LOCATIONS:
Locations (1):
- CADskills HQ, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No